CLINICAL TRIAL: NCT03818334
Title: Use of Post Transplant Cyclophosphamide as Graft Versus Host Disease Prophylaxis in Matched Unrelated Donor Stem Cell Transplantation for Hematological Malignancies, a Prospective Randomized Controlled Trial
Brief Title: Post Transplant Cyclophosphamide in Matched Unrelated Donor Stem Cell Transplantation for Hematological Malignancies
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Andreza Alice Feitosa Ribeiro, Assistant Physician specialist in Hematopoietic Stem Transplantation, Principal Investigator, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SGPP 3549-18
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Bone Marrow Transplant Complications; Graft Versus Host Disease; Infection Viral; Engraft Failure; Immunologic Suppression
Keywords: Bone Marrow Transplantation; Hematological Malignancies; Post-Cy
MeSH Terms: conditions — Graft vs Host Disease; Virus Diseases; Hematologic Neoplasms | interventions — Cyclophosphamide; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Cyclophosphamide (Experimental): Cyclophosphamide 50 mg/Kg on days +3 and +4 AND Calcineurin Inhibitor from day +5 AND Mycofenolate Mofetil from day +5 until day +35
  Interventions: Drug: Cyclophosphamide
- Thymoglobulin (ATG) (Active Comparator): Thymoglobulin (ATG) total dose 5 mg/Kg from day -4 until day -1 AND Calcineurin Inhibitor from day +5 AND Methotrexate on days +1, +3, +6 and +11
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 1000 mg/flask
  Other Names: Cytoxan
  Arms: Post Cyclophosphamide
Drug: ATG — Antihuman T-Lymphocyte Immune Globulin 25 mg/flask
  Other Names: Thymoglobulin
  Arms: Thymoglobulin (ATG)

SUMMARY:
This study aims to evaluate the clinical efficacy of cyclophosphamide in patients receiving a bone marrow graft from a matched unrelated donor in overall survival, progression free survival and cumulative incidence of acute and chronic GvHD. Thirty patients will receive cyclophosphamide while twenty patients will receive antihuman T-lymphocyte immune globulin (ATG).

ELIGIBILITY:
Inclusion Criteria:

* Men and Women of Any Age
* Indication for an HSCT without matched sibling donor
* Have a matched unrelated donor (HLA 10 x 10 or 9 x 10)
* Hematological malignancy

Exclusion Criteria:

* Acute leukemias not in complete response (that is > 5% blast in the bone marrow)
* Chemorefractory lymphoproliferative disease
* Active uncontrolled infection
* HCT-CI > 3
* Severe organic disfunction (heart ejection fraction < 45%, glomerular filtration rate < 50 mL.hour, pulmonary DLCO < 50%)
* Previous allogeneic bone marrow transplantation
* Contraindication to cyclophosphamide or ATG

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  Time to last follow-up or death

SECONDARY OUTCOMES:
Progression free survival | 4 years
  Time until last follow-up, death or disease relapse
Acute Graft Versus Host Disease | 4 years
  Time until acute GvHD development
Chronic Graft Versus Host Disease | 4 years
  Time until chronic GvHD development
Treatment Related Mortality | 4 years
  Time until death related to HSCT complications

OTHER OUTCOMES:
Graft Failure Incidence | 2 years
  ANC < 500/microL after 42 days after graft infusion
Time Until Neutrophil Engraftment | 2 years
  Time to ANC > 500/microL for three consecutive days
Time Until Platelet Engraftment | 2 years
  Time to platelet count > 50,000/microL, without transfusion in the last 7 days
Immunological Reconstitution | Days +60, +100 and +180
  Total lymphocyte count as well as its subsets (CD4, CD8, CD19, CD56)
Days hospitalized | First 100 days after graft infusion
  Days admitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Andreza A Feitosa Ribeiro, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Nelson Hamerschlak, PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospita Israelita Albert Eintein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finke J, Schmoor C, Bethge WA, Ottinger HD, Stelljes M, Zander AR, Volin L, Heim DA, Schwerdtfeger R, Kolbe K, Mayer J, Maertens JA, Linkesch W, Holler E, Koza V, Bornhauser M, Einsele H, Bertz H, Grishina O, Socie G; ATG-Fresenius Trial Group. Prognostic factors affecting outcome after allogeneic transplantation for hematological malignancies from unrelated donors: results from a randomized trial. Biol Blood Marrow Transplant. 2012 Nov;18(11):1716-26. doi: 10.1016/j.bbmt.2012.06.001. Epub 2012 Jun 17. PMID 22713691
- [Background] Bacigalupo A, Lamparelli T, Barisione G, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Sacchi N, van Lint MT, Bosi A; Gruppo Italiano Trapianti Midollo Osseo (GITMO). Thymoglobulin prevents chronic graft-versus-host disease, chronic lung dysfunction, and late transplant-related mortality: long-term follow-up of a randomized trial in patients undergoing unrelated donor transplantation. Biol Blood Marrow Transplant. 2006 May;12(5):560-5. doi: 10.1016/j.bbmt.2005.12.034. PMID 16635791
- [Background] Devillier R, Labopin M, Chevallier P, Ledoux MP, Socie G, Huynh A, Bourhis JH, Cahn JY, Roth-Guepin G, Mufti G, Desmier D, Michallet M, Fegueux N, Ciceri F, Baron F, Blaise D, Nagler A, Mohty M. Impact of antithymocyte globulin doses in reduced intensity conditioning before allogeneic transplantation from matched sibling donor for patients with acute myeloid leukemia: a report from the acute leukemia working party of European group of Bone Marrow Transplantation. Bone Marrow Transplant. 2018 Apr;53(4):431-437. doi: 10.1038/s41409-017-0043-y. Epub 2018 Jan 12. PMID 29330391
- [Background] Saber W, Opie S, Rizzo JD, Zhang MJ, Horowitz MM, Schriber J. Outcomes after matched unrelated donor versus identical sibling hematopoietic cell transplantation in adults with acute myelogenous leukemia. Blood. 2012 Apr 26;119(17):3908-16. doi: 10.1182/blood-2011-09-381699. Epub 2012 Feb 10. PMID 22327226
- [Background] Mehta RS, Saliba RM, Chen J, Rondon G, Hammerstrom AE, Alousi A, Qazilbash M, Bashir Q, Ahmed S, Popat U, Hosing C, Khouri I, Shpall EJ, Champlin RE, Ciurea SO. Post-transplantation cyclophosphamide versus conventional graft-versus-host disease prophylaxis in mismatched unrelated donor haematopoietic cell transplantation. Br J Haematol. 2016 May;173(3):444-55. doi: 10.1111/bjh.13977. Epub 2016 Mar 7. PMID 26947769
- [Background] Rashidi A, Slade M, DiPersio JF, Westervelt P, Vij R, Romee R. Post-transplant high-dose cyclophosphamide after HLA-matched vs haploidentical hematopoietic cell transplantation for AML. Bone Marrow Transplant. 2016 Dec;51(12):1561-1564. doi: 10.1038/bmt.2016.217. Epub 2016 Aug 15. PMID 27526282
- [Background] Moiseev IS, Pirogova OV, Alyanski AL, Babenko EV, Gindina TL, Darskaya EI, Slesarchuk OA, Bondarenko SN, Afanasyev BV. Graft-versus-Host Disease Prophylaxis in Unrelated Peripheral Blood Stem Cell Transplantation with Post-Transplantation Cyclophosphamide, Tacrolimus, and Mycophenolate Mofetil. Biol Blood Marrow Transplant. 2016 Jun;22(6):1037-1042. doi: 10.1016/j.bbmt.2016.03.004. Epub 2016 Mar 10. PMID 26970381
- [Background] Kanakry CG, Bolanos-Meade J, Kasamon YL, Zahurak M, Durakovic N, Furlong T, Mielcarek M, Medeot M, Gojo I, Smith BD, Kanakry JA, Borrello IM, Brodsky RA, Gladstone DE, Huff CA, Matsui WH, Swinnen LJ, Cooke KR, Ambinder RF, Fuchs EJ, de Lima MJ, Andersson BS, Varadhan R, O'Donnell PV, Jones RJ, Luznik L. Low immunosuppressive burden after HLA-matched related or unrelated BMT using posttransplantation cyclophosphamide. Blood. 2017 Mar 9;129(10):1389-1393. doi: 10.1182/blood-2016-09-737825. Epub 2017 Jan 3. PMID 28049637